CLINICAL TRIAL: NCT02217709
Title: Phase 2 Trial of Phenelzine in Non-metastatic Recurrent Prostate Cancer
Brief Title: Phenelzine Sulfate in Treating Patients With Non-metastatic Recurrent Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4P-14-1; NCI-2014-01791 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HS-14-00331; 4P-14-1 (Other: USC Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2014-08-13; First posted 2014-08-15 (Estimated); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Adenocarcinoma of the Prostate; Recurrent Prostate Cancer; Stage I Prostate Cancer; Stage IIA Prostate Cancer; Stage IIB Prostate Cancer; Stage III Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Phenelzine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (phenelzine sulfate) (Experimental): Patients receive phenelzine sulfate 30 mg by mouth (PO) twice daily (BID) (starting dose of 15 mg daily escalated to 30 mg BID over 16 plus or minus 5 days). Patients who have been treated at 30 mg BID for over 3 cycles with resolution of any and all toxicities to grade < or = 1 may increase the dose to a maximum of 45 mg BID at the discretion of the treating investigator. Treatment may continue in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: phenelzine sulfate; Other: laboratory biomarker analysis; Other: questionnaire administration

INTERVENTIONS:
Drug: phenelzine sulfate — Given by mouth
  Other Names: Nardil
Other: laboratory biomarker analysis — Correlative studies
Other: questionnaire administration — Ancillary studies

SUMMARY:
This phase II trial studies phenelzine sulfate in treating patients with prostate cancer that has not spread to other parts of the body and has come back. Phenelzine sulfate is a type of antidepressant that works by decreasing the amount of a protein called monoamine oxidase (MAO). MAO drugs may have an anticancer effect in prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the proportion of patients with biochemical recurrent prostate cancer (BCR-PC) treated with phenelzine (phenelzine sulfate) who achieve a prostate-specific antigen (PSA) decline of >= 50% from baseline.

SECONDARY OBJECTIVES:

I. To monitor potential toxicities and/or beneficial effects on quality of life of phenelzine in prostate cancer patients.

II. To assess time to radiographic disease progression for patients with recurrent prostate cancer treated with phenelzine.

III. To collect blood and other samples to study the relationship between MAO activity and prostate cancer.

OUTLINE:

Patients receive phenelzine sulfate 30 mg by mouth (PO) twice daily (BID) (starting dose of 15 mg daily escalated to 30 mg BID over 16 plus or minus 5 days). Patients who have been treated at 30 mg BID for over 3 cycles with resolution of any and all toxicities to grade < or = 1 may increase the dose to a maximum of 45 mg BID at the discretion of the treating investigator. Treatment may continue in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate
* Recurrent prostate cancer following primary therapy as defined by:

  * Post-radical prostatectomy: Any PSA >= 0.4 ng/ml
  * Post-primary radiotherapy: PSA >= 2 ng/ml above a post-radiotherapy nadir
  * Post-primary androgen-deprivation therapy: A confirmed rise of PSA >= 2 ng/ml above a post-therapy nadir
* For patients with non-castrate levels of circulating androgen levels (testosterone >= 50 g/dl)

  * PSA levels should be increasing on at least two occasions >= 1 week apart
  * Patients should not be considered candidates for radiation therapy
* For patients with castrate levels of circulating androgen levels (testosterone < 50 ng/dl):

  * PSA levels must be >= 0.4 ng/ml (if history of radical prostatectomy) or >= 2 ng/ml (if history of non-surgical primary treatment) and found to be increasing on at least two occasions >= 1 week apart
* At least 4 weeks must have elapsed since any changes to hormonal therapy, including at least 4 weeks since flutamide and at least 6 weeks since bicalutamide, nilutamide, or enzalutamide
* No evidence of metastatic cancer on imaging including a bone scan and computed tomography (CT) scan of chest/abdomen/pelvis
* Able to understand and adhere to dietary and medication restrictions as recommended for the safe use of phenelzine
* Men with child bearing potential are required to use an effective means of contraception
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 x upper limit of normal (ULN) except in cases of benign isolated hyperbilirubinemia such as Gilbert's syndrome.
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SPGT]) =< 2.5 x ULN
* Creatinine =< 1.5 x ULN

Exclusion Criteria:

* Uncontrolled hypertension despite appropriate medical therapy (blood pressure [BP] greater than 160 mmHg systolic and 90 mmHg diastolic at 2 separate measurements no more than 60 minutes apart during the screening visit); Note: patients may be rescreened after adjustment of antihypertensive medications
* Known prior history of mania or major psychiatric illness (schizophrenia, bipolar disorder, severe major depression requiring hospitalization, etc.)
* Concurrent use of medications contra-indicated due to potential interactions with phenelzine
* Inability to comply with dietary restrictions for foods, supplements, and medications with potential for adverse interactions with phenelzine or to otherwise cooperate fully with the investigator and study personnel
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to phenelzine or other monoamine oxidase inhibitors
* Patients may not be receiving any other investigational agents
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-09-08 (Actual); Primary Completion 2020-06-29 (Actual); Study Completion 2020-06-29 (Actual)

PRIMARY OUTCOMES:
Occurrence of PSA decline to >= 50% from baseline following at least 12 weeks of treatment with phenelzine sulfate | Baseline to up to 12 months
  Assessed independently in two groups of patients defined according to circulating androgen levels as: non-castrate and castrate.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Gross, MD, Principal Investigator — University of Southern California; Jean C. Shih, PhD, Principal Investigator — University of Southern California
Locations (4):
- United States (4):
  - USC Norris Westside Cancer Center, Beverly Hills, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Keck Medical Center of USC Pasadena, Pasadena, California